CLINICAL TRIAL: NCT01958073
Title: Vaginal Estrogen for the Prevention of Recurrent Urinary Tract Infection in Postmenopausal Women: A Randomized Clinical Trial
Brief Title: Vaginal Estrogen for the Prevention of Recurrent Urinary Tract Infection in Postmenopausal Women
Acronym: VESPR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Urogynecologic Society (Other); NYU Langone Health (Other)
Responsible Party: Principal Investigator, Kimberly Ferrante, MD, Female Pelvic Medicine and Reconstructive Surgery Attending, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 130403
Record Dates: First submitted 2013-03-27; First posted 2013-10-08 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Recurrent Urinary Tract Infection; Postmenopausal; Vaginal Estrogen
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conjugated Estrogen Vaginal Cream (Experimental): Conjugated estrogen vaginal cream 0.5g per vagina 2 times weekly
  Interventions: Drug: Conjugated Estrogen Vaginal Cream
- Estradiol Ring (Experimental): Estradiol Ring per vagina every 3 months
  Interventions: Drug: Estradiol Ring
- Placebo (Placebo Comparator): Per vagina
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Conjugated Estrogen Vaginal Cream
  Arms: Conjugated Estrogen Vaginal Cream
Drug: Estradiol Ring
  Arms: Estradiol Ring
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators would like to know if the use of vaginally applied estrogen can prevent the problem of repeated urinary tract infections (UTI) in women who have gone through menopause. The investigators will use two forms of vaginal estrogen that are available by prescription (a ring and a cream) and compare their efficacy to that of a placebo (without any active ingredient). The investigators are going to look at if the vaginal estrogen can prevent UTIs altogether and also the number of UTIs each group experiences over a 6 month period. After 6 months, all subjects will receive vaginal estrogen and the women on the non-active treatment will be able to choose whether they would like to use either the estrogen ring or cream. The investigators will then be able to compare the number of UTIs on and off active vaginal estrogen treatment within those subjects who started on the placebo. The investigators are also going to look at quality of life before and during treatment using questionnaires and whether subjects stop using the treatments or do not use them as directed (compliance).

DETAILED DESCRIPTION:
This was an investigator-initiated, multicenter, single-blind, randomized placebo-controlled trial of vaginal estrogen (delivered by estradiol ring or conjugated estrogen cream) compared to placebo cream. This study was conducted by the Divisions of Female Pelvic Medicine and Reconstructive Surgery at three academic institutions.

Potential participants were recruited from women receiving care for rUTIs in the clinics of each institution. Women were postmenopausal as defined by amenorrhea for >12 months, history of bilateral salpingoophrectomy, or in patients with prior hysterectomy defined as menopausal symptoms for >1 year or age >55. Participants had documented rUTI (three or more in one year or two in six months) by positive urine culture. Participants were excluded if they had undergone urologic surgery within three months of screening or planned surgery within one year of screening, had the diagnosis of painful bladder syndrome, history of UTI requiring the use of intravenous antibiotics or one oral antibiotic available for treatment based on allergies and resistance profiles, known etiology of infections (e.g. urologic stones, fistulas, fecal incontinence, catheterization or poorly controlled diabetes), urothelial cancer, or actively treated estrogen sensitive tumor. Participant enrollment was deferred in the setting of undiagnosed hematuria or vaginal bleeding, but enrollment could occur after negative workup for malignancy. Participants deferred enrollment if they used vaginal androgens, estrogens or progestins within six months or if they used medications or supplements known to prevent UTI (e.g. cranberry products, D mannose, prophylactic antibiotics, methenamine hippurate) within three months of enrollment, but could enroll after washout. Those with a remote history of estrogen-sensitive tumor required approval by her oncologist or primary care physician.

Participants were initially randomized to receive either vaginal estrogen (via estradiol ring or conjugated estrogen cream) or placebo cream in a 1:1:1 fashion and were told that there were placebo and vaginal estrogen arms, but were unaware that there was not a placebo ring. Participants were randomized to either conjugated estrogen cream at a strength of 0.625 mg/g dosed at 0.5g (0.312 mg) twice a week, estradiol ring containing 2mg of estradiol placed vaginally every three months by study personnel, or placebo cream which was an over-the-counter lubricant containing mineral oil, petrolatum, ceresin and paraffin dosed at 0.5g twice a week. If participants in any arm developed three UTI in the six-month treatment period, they were unblinded. If on placebo, they were provided active study drug or if they were in the vaginal estrogen arm, they were treated according to the provider's clinical practice and their outcomes recorded for the remainder of the study. The primary outcome of occurrence of UTI was assessed at six months or the end of study blinding, whichever occurred first. In order to improve recruitment and assess long-term compliance, satisfaction and efficacy, we offered open label use of estradiol ring or conjugated estrogen cream after unblinding until month 12 of the study.

Clean-catch urine cultures were collected when participants were symptomatic: fever (>38 degrees C), urgency, frequency, dysuria or suprapubic tenderness. Women were asked to have all urine labs done at the parent site as per standard clinical practice. The primary outcome of the study was the presence of a UTI in the randomized six months. We also assessed rates of UTI over the course of the 12-month study in all participants as-treated. Quality of life (QOL) questionnaires were administered at baseline, six months or unblinding, and 12 months. Questionnaires included the Pelvic Floor Distress Inventory (PFDI-20), Pelvic Floor Impact Questionnaire (PFIQ-7), Medical, Epidemiologic, and Social Aspects of Aging Questionnaire (MESA), Female Sexual Function Index (FSFI) and Patient Satisfaction Questionnaire (PSQ), Global Perception of Improvement (GPI) and Estimated Percent Improvement (EPI) rating scales. Baseline medical history and concomitant pelvic medicine diagnoses were also collected. Participants using a cream treatment were asked to keep medication diaries and return tubes for weighing at months three, six, nine and 12. Adherence was defined as presence of the estrogen ring or tube weights within 20% of expected at follow up visits. In addition, before unblinding, the participants were asked whether they believed they were on active treatment, placebo, or were unsure.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal status as defined by amenorrhea for >12 months, OR history of bilateral salpingoophrectomy, OR if the patient has had a hysterectomy defined by menopausal symptoms for >1 year OR age >55
2. Documented recurrent UTIs (3 or more in the last year or 2 or more in the last 6 months)- one UTI must be documented by culture, others may be documented by urinalysis
3. Ability to provide informed consent

Exclusion Criteria:

1. Use of any investigational drug or device within thirty days of screening
2. Urologic surgery within the past 3 months of screening or plan for surgery within one year of screening
3. Diagnosis of Interstitial Cystitis/painful bladder syndrome
4. History of urinary tract infections which require the use of IV antibiotics or where only one oral antibiotic is available for treatment, or where the risk of treatment with vaginal estrogen only is deemed unacceptable by the principle investigator secondary to the severity of prior urinary tract infections
5. Known etiology of infection such as, but not limited to: kidney or bladder stones, enterovaginal/vesical fistula, fecal incontinence, intermittent catheterization, indwelling catheter, poorly controlled diabetes
6. Urothelial cancer
7. Actively treated estrogen sensitive tumor (breast or endometrial cancer)
8. Undiagnosed vaginal bleeding
9. Inability to use a vaginal ring (secondary to advanced prolapse or shortened vaginal length)
10. Any medical reason the investigator deems incompatible with treatment with vaginal estrogen
11. Prolapse requiring pessary use

Deferral Criteria

1. Undiagnosed hematuria - may enroll after malignancy is ruled out
2. Use of a progestin containing intrauterine device or use of any vaginal androgens, estrogens or progestins within 3 months of enrollment - may enroll after wash out
3. Use of drugs/supplements known to prevent UTIs (ie cranberry products, prophylactic antibiotics, methenamine hippurate) 1 month prior to enrollment - may enroll after wash out if still meets inclusion criteria.
4. History of estrogen sensitive tumor (breast or endometrial cancer) - requires approval by the subject's primary oncologist or primary care physician

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - New York University Langone Medical Center, New York, New York

REFERENCES:
- [Derived] Ferrante KL, Wasenda EJ, Jung CE, Adams-Piper ER, Lukacz ES. Vaginal Estrogen for the Prevention of Recurrent Urinary Tract Infection in Postmenopausal Women: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):112-117. doi: 10.1097/SPV.0000000000000749. PMID 31232721

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the start of the study we began with the intent of 3 groups for analysis, separating the two forms of vaginal estrogen into separate groups and comparing them to a placebo group. Due to difficulties with recruitment, our protocol was amended so that the two vaginal estrogen groups were combined to one vaginal estrogen group compared to placebo.
Groups:
- Conjugated Estrogen Vaginal Cream; Vaginal Cream Open Label: Conjugated estrogen vaginal cream 0.5g per vagina 2 times weekly
  Conjugated Estrogen Vaginal Cream
- Estradiol Ring; Estradiol Ring Open Label: Estradiol Ring per vagina every 3 months
  Estradiol Ring
- Placebo: Per vagina 0.5g 2 times weekly
  Placebo
Period: Randomized Period
Arm/Group | Conjugated Estrogen Vaginal Cream | Estradiol Ring | Placebo | Vaginal Cream Open Label | Estradiol Ring Open Label
Started | 9 | 9 | 17 | 0 | 0
Completed | 7 | 8 | 11 | 0 | 0
Not Completed | 2 | 1 | 6 | 0 | 0
Period: Open Label Period
Arm/Group | Conjugated Estrogen Vaginal Cream | Estradiol Ring | Placebo | Vaginal Cream Open Label | Estradiol Ring Open Label
Started | 0 | 0 | 0 | 5 | 17
Completed | 0 | 0 | 0 | 5 | 17
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: At the start of the study we began with the intent of 3 groups for analysis, separating the two forms of vaginal estrogen into separate groups and comparing them to a placebo group. Due to difficulties with recruitment, our protocol was amended so that the two vaginal estrogen groups were combined to one vaginal estrogen group compared to placebo.
Groups:
- Vaginal Estrogen: Conjugated estrogen vaginal cream 0.5g per vagina 2 times weekly
  OR
  Estradiol Ring per vagina every 3 months
- Total: Total of all reporting groups
Arm/Group | Placebo | Vaginal Estrogen | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.47) | 72.8 (8.4) | 70.15 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 34
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.41 (7.09) | 30.33 (9.21) | 29.37 (8.15)
Number of UTIs in prior 12 months [Count of Participants; unit: Participants]
  2 | 6 | 7 | 13
  3 | 7 | 9 | 16
  4 | 2 | 1 | 3
  5 | 1 | 1 | 2
  6 | 1 | 0 | 1
Smoking [Count of Participants; unit: Participants]
  Current | 1 | 1 | 2
  Former | 8 | 7 | 15
  Never | 8 | 10 | 18
Marital Status [Count of Participants; unit: Participants]
  Single | 0 | 3 | 3
  Married | 6 | 5 | 11
  Divorced/Separated | 7 | 2 | 9
  Widowed | 3 | 8 | 11
  Other | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  Less than High School | 0 | 1 | 1
  High School/GED | 5 | 4 | 9
  Associates Degree | 3 | 4 | 7
  4 year college | 5 | 5 | 10
  Graduate School | 4 | 4 | 8
Caffeine use [Count of Participants; unit: Participants] | 14 | 14 | 28
Prior Pelvic Surgery [Count of Participants; unit: Participants] | 9 | 13 | 22
Prior Vaginal Estrogen [Count of Participants; unit: Participants] | 4 | 1 | 5
Hormone Replacement Therapy [Count of Participants; unit: Participants]
  Never | 10 | 6 | 16
  Past | 5 | 10 | 15
  Current | 2 | 1 | 3
Diabetes [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of UTI During Randomization
Description: The primary purpose of this study is to assess the efficacy of vaginal estrogen versus placebo at 6 months on the prevention of urinary tract infections (UTI) in postmenopausal women with history of recurrent UTI.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Count of Participants; unit: Participants
Groups:
- Vaginal Estrogen: Conjugated Estrogen Vaginal Cream
  OR
  Estradiol Ring
- Placebo: Per vagina
  Placebo
Arm/Group | Vaginal Estrogen | Placebo
Number analyzed (Participants) | 15 | 11
Participants | 8 | 10

2. Secondary Outcome: Rates of UTI in Both Randomization Period and Within Placebo When Changed to Open Label Estrogen
Description: 1. To assess overall rates of UTI over 6 months in postmenopausal women with history of recurrent UTI receiving vaginal estrogen (ring or cream).
  2. To compare rates of UTI between 6 and 12 months of those subjects initially randomized to placebo.
Time Frame: Assessed at 6 months for 'a'; assessed over 12 months for 'b'
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo During Randomization: Per vagina 0.5g 2 times weekly
  Placebo
- Initial Placebo to Open Label Vaginal Estrogen: Those participants initially randomized to placebo, during the period when they went on open label vaginal estrogen.
Arm/Group | Placebo During Randomization | Vaginal Estrogen | Initial Placebo to Open Label Vaginal Estrogen
Number analyzed (Participants) | 11 | 15 | 10
Participants
  No UTI | 1 | 8 | 7
  1 UTI | 7 | 3 | 2
  2 UTI | 2 | 4 | 1
  3 UTI | 1 | 0 | 0

3. Secondary Outcome: Quality of Life Questionnaire: Female Sexual Function Index
Description: To assess the impact of treatment of recurrent UTI with vaginal estrogen on quality of life at 6 months in postmenopausal women with history of recurrent UTI. Female Sexual Function Index. Scale range 2-95. Lower score corresponds to worse functioning.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaginal Estrogen
Number analyzed (Participants) | 11 | 15
score on a scale | 43.45 (27.83) | 30.64 (29.38)

4. Secondary Outcome: Compliance During Randomization
Description: To assess compliance with vaginal estrogen (ring or cream) treatment at 6 months in postmenopausal women with history of recurrent UTI.
Time Frame: 6 months of the randomized period
Population: as treated, we did not collect data from the placebo group; although vaginal estrogen groups were combined in a protocol amendment for the primary outcome, they were not combined for this secondary outcome looking at compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Conjugated Estrogen Vaginal Cream | Estradiol Ring
Number analyzed (Participants) | 7 | 8
Participants | 4 | 8

5. Secondary Outcome: Occurrence of UTI in Those Compliant With Treatment During Randomization
Description: To assess efficacy of vaginal estrogen at 6 months in those compliant with treatment.
Time Frame: 6 months of the randomized period
Population: as treated; although vaginal estrogen groups were combined in a protocol amendment for the primary outcome, they were not combined for this secondary outcome looking at compliance. Compliance was not assessed in placebo which was used as a comparator group for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Conjugated Estrogen Vaginal Cream | Estradiol Ring | Placebo
Number analyzed (Participants) | 4 | 8 | 11
Participants | 3 | 5 | 10

6. Secondary Outcome: Quality of Life Questionnaire: MESA I
Description: To assess the impact of treatment of recurrent UTI with vaginal estrogen on quality of life at 6 months in postmenopausal women with history of recurrent UTI. Medical, Epidemiologic, and Social Aspects of Aging Questionnaire (MESA) urinary incontinence questionnaire: stress urinary incontinence subscale. Subscale range 0-27. A higher score indicated more frequent symptoms.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaginal Estrogen
Number analyzed (Participants) | 11 | 15
score on a scale | 7.00 (7.27) | 9.86 (6.93)

7. Secondary Outcome: Quality of Life Questionnaire: MESA II
Description: To assess the impact of treatment of recurrent UTI with vaginal estrogen on quality of life at 6 months in postmenopausal women with history of recurrent UTI. Medical, Epidemiologic, and Social Aspects of Aging Questionnaire (MESA) urinary incontinence questionnaire: urgency urinary incontinence subscale. Subscale range 0-18. High score indicates more frequent symptoms.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaginal Estrogen
Number analyzed (Participants) | 11 | 15
score on a scale | 4.82 (5.76) | 4.79 (3.21)

8. Secondary Outcome: Quality of Life Questionnaire: Pelvic Floor Disability Index
Description: To assess the impact of treatment of recurrent UTI with vaginal estrogen on quality of life at 6 months in postmenopausal women with history of recurrent UTI. Pelvic Floor Disability Index. Scale range 0-100. Higher score corresponds to increased bother.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaginal Estrogen
Number analyzed (Participants) | 11 | 15
score on a scale | 65.88 (56.29) | 55.53 (31.76)

9. Secondary Outcome: Quality of Life Questionnaire: Pelvic Floor Impact Questionnaire
Description: To assess the impact of treatment of recurrent UTI with vaginal estrogen on quality of life at 6 months in postmenopausal women with history of recurrent UTI. Pelvic Floor Impact Questionnaire. Scale range 0-300. Higher score corresponds to increasing bother.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaginal Estrogen
Number analyzed (Participants) | 11 | 15
score on a scale | 22.08 (44.01) | 9.86 (14.88)

10. Secondary Outcome: Quality of Life Questionnaire: Estimated Percentage of Improvement
Description: To assess the impact of treatment of recurrent UTI with vaginal estrogen on quality of life at 6 months in postmenopausal women with history of recurrent UTI. Estimated Percentage of Improvement. Scale range 0-100. Higher score corresponds to more improvement.
Time Frame: 6 months of the randomized period
Population: As treated. Vaginal estrogen groups were combined due to a protocol amendment.
Measure: Mean (Standard Deviation); unit: percentage of improvement
Arm/Group | Placebo | Vaginal Estrogen
Number analyzed (Participants) | 11 | 15
percentage of improvement | 33.00 (35.48) | 74.64 (25.83)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 1 year after start of study participation
Groups:
- Vaginal Estrogen Cream Randomization; Vaginal Estrogen Cream Open Label: Conjugated estrogen vaginal cream 0.5g per vagina 2 times weekly
- Vaginal Estrogen Ring Randomization; Vaginal Estrogen Ring Open Label: Estradiol Ring per vagina every 3 months
Arm/Group | Placebo | Vaginal Estrogen Cream Randomization | Vaginal Estrogen Ring Randomization | Vaginal Estrogen Cream Open Label | Vaginal Estrogen Ring Open Label
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/9 | 0/9 | 0/5 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/9 | 0/9 | 0/5 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/9 | 0/9 | 0/5 | 0/17

LIMITATIONS AND CAVEATS:
Difficult recruitment requiring several modifications to the study design, single-blind nature of the trial, underpowered for secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT01958073/Prot_SAP_000.pdf